CLINICAL TRIAL: NCT01470118
Title: A Study to Evaluate the Duration of LASTACAFT® in Acute Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMA-LAS-011-001
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-01

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine; Ophthalmic Solutions; Olopatadine Hydrochloride; Dextrans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LASTACAFT® (alcaftadine 0.25%) (Active Comparator): One drop of alcaftadine 0.25% ophthalmic solution instilled in each eye at Day 0 and Day 14.
  Interventions: Drug: alcaftadine 0.25% ophthalmic solution
- Pataday™ (olopatadine 0.2%) (Active Comparator): One drop of olopatadine 0.2% ophthalmic solution instilled in each eye at Day 0 and Day 14.
  Interventions: Drug: olopatadine 0.2% ophthalmic solution
- Placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%) (Placebo Comparator): One drop of placebo instilled in each eye at Day 0 and Day 14.
  Interventions: Drug: dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%

INTERVENTIONS:
Drug: alcaftadine 0.25% ophthalmic solution — One drop of alcaftadine 0.25% ophthalmic solution instilled in each eye at Day 0 and Day 14.
  Other Names: LASTACAFT®
  Arms: LASTACAFT® (alcaftadine 0.25%)
Drug: olopatadine 0.2% ophthalmic solution — One drop of olopatadine 0.2% ophthalmic solution instilled in each eye at Day 0 and Day 14.
  Other Names: Pataday™
  Arms: Pataday™ (olopatadine 0.2%)
Drug: dextran 70 0.1%/hydroxypropyl methylcellulose 0.3% — One drop of placebo instilled in each eye at Day 0 and Day 14.
  Other Names: Tears Naturale® II Artificial Tears
  Arms: Placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%)

SUMMARY:
This study will evaluate the duration of action of LASTACAFT® and Pataday™ as compared to artificial tears (placebo) in the prevention of ocular itching associated with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of eye allergies within the past 24 months
* Willing to not wear contact lenses at least 72 hours prior to the study start and during the study period

Exclusion Criteria:

* Current eye infection
* Eye surgery within 3 months or vision correction surgery within 6 months
* Any planned surgery during the study or 30 days after the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] McLaurin EB, Marsico NP, Ackerman SL, Ciolino JB, Williams JM, Villanueva L, Hollander DA. Ocular itch relief with alcaftadine 0.25% versus olopatadine 0.2% in allergic conjunctivitis: pooled analysis of two multicenter randomized clinical trials. Adv Ther. 2014 Oct;31(10):1059-71. doi: 10.1007/s12325-014-0155-3. Epub 2014 Sep 27. PMID 25260889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Started | 43 | 43 | 41
Completed | 38 | 38 | 39
Not Completed | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%) | Total
Number analyzed (Participants) | 43 | 43 | 41 | 127
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (12.44) | 37.0 (14.84) | 39.3 (12.31) | 38.5 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 28 | 92
  Male | 12 | 10 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Evaluated by the Subject at 3, 5, and 7 Minutes Post Challenge on Day 0 at Hour 16
Description: Ocular itching evaluated by the subject at 3, 5, and 7 minutes post challenge on Day 0 (Visit 3) at hour 16. Subjects scored their ocular itching on a numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less itching.
Time Frame: Day 0 Hour 16
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  3 Minutes | 0.62 (0.716) | 1.01 (0.8211) | 2.14 (0.864)
  5 Minutes | 0.93 (0.789) | 1.13 (0.852) | 2.35 (0.759)
  7 Minutes | 1.07 (0.830) | 1.12 (0.824) | 2.20 (0.888)

2. Secondary Outcome: Conjunctival Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Conjunctival redness evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Investigators scored conjunctival redness on a numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less conjunctival redness.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 1.74 (0.612) | 1.78 (0.709) | 2.08 (0.605)
  15 Minutes | 2.01 (0.672) | 2.01 (0.805) | 2.22 (0.671)
  20 Minutes | 1.99 (0.652) | 1.92 (0.870) | 2.20 (0.691)

3. Secondary Outcome: Ciliary Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Ciliary redness evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Investigators scored ciliary redness on a numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less ciliary redness.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 1.36 (0.730) | 1.47 (0.773) | 1.83 (0.764)
  15 Minutes | 1.64 (0.805) | 1.67 (0.901) | 2.00 (0.772)
  20 Minutes | 1.67 (0.754) | 1.65 (0.909) | 1.94 (0.844)

4. Secondary Outcome: Episcleral Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Episcleral redness evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Investigators scored episcleral redness on a numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less episcleral redness.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 1.65 (0.667) | 1.56 (0.827) | 2.01 (0.682)
  15 Minutes | 1.95 (0.649) | 1.82 (0.924) | 2.15 (0.727)
  20 Minutes | 1.91 (0.645) | 1.79 (0.960) | 2.13 (0.718)

5. Secondary Outcome: Chemosis Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Chemosis evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Investigators scored chemosis on a numeric analog scale ranging from 0=None to 4=Severe (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less chemosis.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 0.90 (0.392) | 0.97 (0.479) | 1.15 (0.505)
  15 Minutes | 1.03 (0.403) | 1.09 (0.616) | 1.34 (0.668)
  20 Minutes | 1.14 (0.457) | 1.13 (0.677) | 1.42 (0.742)

6. Secondary Outcome: Eyelid Swelling Evaluated by the Subject at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Eyelid swelling evaluated by the subject at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Subjects scored eyelid swelling on a numeric analog 4-point scale ranging from 0=None to 3=Severe. For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less lid swelling.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 0.4 (0.62) | 0.4 (0.51) | 1.0 (0.75)
  15 Minutes | 0.5 (0.66) | 0.6 (0.74) | 1.0 (0.88)
  20 Minutes | 0.6 (0.65) | 0.6 (0.77) | 1.1 (0.87)

7. Secondary Outcome: Tearing Evaluated by the Subject at 7, 15, and 20 Minutes Post Challenge on Day 14 at Hour 24
Description: Tearing evaluated by the subject at 7, 15, and 20 minutes post challenge on Day 14 (Visit 4) at hour 24. Subjects scored tearing on a 5-point numeric analog scale ranging from 0=None/Normal to 4=Very Severe. For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less tearing.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  7 Minutes | 0.3 (0.49) | 0.4 (0.81) | 1.0 (0.91)
  15 Minutes | 0.5 (0.62) | 0.6 (0.93) | 0.9 (0.87)
  20 Minutes | 0.5 (0.60) | 0.6 (1.03) | 0.8 (0.86)

8. Primary Outcome: Ocular Itching Evaluated by the Subject at 3, 5, and 7 Minutes Post Challenge on Day 14 at Hour 24
Description: Ocular itching evaluated by the subject at 3, 5, and 7 minutes post challenge on Day 14 (Visit 4) at hour 24. Subjects scored their ocular itching on a numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments were allowed). For each subject, the score for both eyes was averaged (i.e., one score per subject). A lower score was indicative of less itching.
Time Frame: Day 14 Hour 24
Population: Intent-to-Treat: All randomized subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 43 | 43 | 41
Scores on a Scale
  3 Minutes | 0.64 (0.807) | 0.97 (0.771) | 2.27 (0.846)
  5 Minutes | 0.84 (0.851) | 1.16 (0.886) | 2.19 (0.897)
  7 Minutes | 0.93 (0.911) | 1.01 (0.932) | 1.96 (1.068)

ADVERSE EVENTS:
Description: The Safety Population was defined as all randomized subjects who received at least one dose of study treatment and was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | LASTACAFT® (Alcaftadine 0.25%) | Pataday™ (Olopatadine 0.2%) | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo